CLINICAL TRIAL: NCT07282353
Title: A Randomized, Double-Blind, Placebo-controlled, Phase III Study to Evaluate the Efficacy and Safety of CS0159 in Patients With Primary Biliary Cholangitis (PBC) With Inadequate Response or Intolerance to Ursodeoxycholic Acid (UDCA)
Brief Title: A Study of CS0159 in Patients With PBC With Inadequate Response or Intolerance to UDCA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cascade Pharmaceuticals, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS0159-PBC-CN-III-07
Record Dates: First submitted 2025-11-21; First posted 2025-12-15 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 mg CS0159 (Experimental): Take 4mg of CS0159 QD for 52 weeks.
  Interventions: Drug: 2mg CS0159
- placebo (Placebo Comparator): Take placebo QD for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 2mg CS0159 — Oral QD
  Arms: 4 mg CS0159
Drug: Placebo — Oral QD
  Arms: placebo

SUMMARY:
A Randomized, Double-Blind, Placebo-controlled, Phase III Study to Evaluate the Efficacy and Safety of CS0159 in Patients with Primary Biliary Cholangitis (PBC) with inadequate response or intolerance to ursodeoxycholic acid (UDCA).

DETAILED DESCRIPTION:
This is an multicenter, randomized, double-blind, placebo-controlled, parallel-group study that evaluates the efficacy and safety of CS0159 in patients with PBC who have inadequate response or intolerance to ursodeoxycholic acid (UDCA). Approximately 135 participants will be randomized in a 2:1 ratio to receive CS0159 (4 mg) or placebo, once daily, for a maximum of 52 weeks. When applicable, study participants should continue their pre-study dose of UDCA.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated) and any authorizations required by local law;
2. When signing ICF age ≥18 years ≤75 years, male or female;
3. Meets the diagnostic criteria of PBC, based on any two of the following criteria:

   1. History of ALP above 1.0× ULN for at least 6 months
   2. Positive antimitochondrial antibody (AMA) titer (>1:40 on immunofluorescence or M2 positive by ELISA) or positive PBC- specific antinuclear antibody (ANA) (either SP100 or GP210 positive)
   3. Documented liver biopsy results consistent with PBC;
4. UDCA≥6 months before randomization and a stable dose ≥3 months after the efficacy was poor [meeting inclusion criteria (5)a], or UDCA was not tolerated, and stop taking UDCA (no UDCA use for ≥3 months before randomization);
5. Central laboratory parameters measured at screening period meet the following criteria:

   1. ALP ≥1.67× ULN
   2. ALT≤5× ULN
   3. AST ≤5× ULN
   4. TB <2× ULN
   5. Estimated glomerular filtration rate (eGFR) > 60mL/min/1.73m2 (calculated by CKD-EPI equation)
   6. INR ≤ 1.0× ULN. For participants on anticoagulation therapy, INR must be maintained in the range required for prophylaxis for their specific disease
   7. Platelet count ≥ 150× 109/μL (No thrombocytopenia-related treatment within the past two weeks)
   8. Albumin> 35g/L
   9. White blood cells count (WBC) >3×109/L
   10. Absolute neutrophil count (ANC) >1.5×109/L
   11. Hemoglobin A1c (HbA1c) ≤9.0%;
6. Females of reproductive potential must use at least 1 barrier contraceptive and a second effective birth control method during the study and for at least 90 days after the last dose. Male participants who are sexually active with female partners of reproductive potential must use barrier contraception, and their female partners must use a second effective birth control method during the study and for at least 90 days after the last dose.

   -

Exclusion Criteria:

1. Previous exposure to CS0159;
2. History of allergy to the CS0159 or its excipients or drugs of similar chemical classes;
3. Advanced PBC as defined by the Rotterdam criteria (albumin<1.0×LLN AND TB >1.0× ULN);
4. Patients who have had clinically significant complications of hepatic cirrhosis with clinically significant portal hypertension (CSPH), including the following:

   1. History of liver transplantation, current placement on a liver transplant list, current MELD -Na score ≥ 12;
   2. History of confirmed esophagogastric variceal bleeding;
   3. Clinically significant ascites requiring intervention, such as sodium restriction, diuretic therapy, or therapeutic paracentesis;
   4. Any secondary complications resulting from clinically significant ascites, such as spontaneous bacterial peritonitis, hepatorenal syndrome, or hepatic hydrothorax;
   5. Hepatic encephalopathy requiring drug therapy;
   6. Portopulmonary hypertension and/or hepatopulmonary syndrome;
   7. Hepatocellular carcinoma;
5. Other concomitant liver disease including:

   1. Autoimmune hepatitis (AIH) (simplified AIH diagnostic score >6), PBC-AIH overlap syndrome, or overlap with other autoimmune liver diseases
   2. Positive HBsAg or positive HCV RNA (tested for in case of known cured HCV infection or positive HCV Ab at screening)
   3. Primary sclerosing cholangitis (PSC)
   4. History or clinical evidence of Alcoholic liver disease (ALD)
   5. Biopsy confirmed Non-alcoholic steatohepatitis (NASH)
   6. Gilbert's Syndrome
   7. History or evidence of alpha-1 antitrypsin deficiency
   8. Liver stiffness measured by transient elastography (TE) > 16.9 Kpa;
6. Patient has a positive test for HIV at screening, or active syphilis [defined as positive Treponema pallidum antibody (TP Ab) and a rapid plasma reagin (RPR) card test titer ≥1:8; for low titers (e.g., 1:1 or 1:2), clinical judgment is required to determine if it is active syphilis];
7. Administration of the following medications are prohibited as specified below:

   1. Use of medications, food, and drinks (e.g., grapefruit juice) that are strong or moderate CYP3A4 inhibitors or inducers within 14 days before randomization;
   2. Use of P-glycoprotein (P-gp) substrate drugs within 14 days before randomization;
   3. 2 months prior to randomization: fibrates, glitazones, seladelpar and elafibranor.
   4. 3 months prior to randomization: obeticholic acid (OCA), azathioprine, colchicine, cyclosporine, methotrexate, mycophenolate, pentoxifylline, systemic corticosteroids and budesonide (˃2 weeks); potentially hepatotoxic drugs (including α-methyl-dopa, sodium valproic acid isoniazid, or nitrofurantoin).
   5. Patients with systemic treatment for pruritus (e.g., with bile acid sequestrants [BAS]) within 3 months prior to randomization.
   6. 12 months prior to randomization: antibodies or immunotherapy directed against ILs or other cytokines or chemokines;
8. Medical conditions that may cause non-hepatic increases in ALP (e.g., paget's disease);
9. Patients with severe arrhythmia, or a QTcF interval corrected by Fridericia's formula ≥450 ms (males) or ≥470 ms (females) at screening [Fridericia's formula: QTcF=QT/(RR^0.33)];
10. History or presence of any disease or condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs including bile salt metabolism in the large intestine, eg, inflammatory bowel disease, prior or planned (during the study period) bariatric surgery (such as gastroplasty, roux-en-Y gastric bypass);
11. History of malignancy (except for those with a disease-free survival of ≥5 years) or currently under evaluation for malignancy; except for cured squamous or non-invasive skin basal cell carcinoma and cervical carcinoma in situ;
12. Drug abuse or heavy alcohol use from 12 months prior to randomization throughout the entire clinical study period. Heavy alcohol use is defined as an average weekly alcohol consumption of more than approximately 7 standard drinks for females and more than approximately 14 standard drinks for males. One standard drink is defined as any beverage containing 14g of pure alcohol, such as 12 oz/360 mL of beer (5% alcohol), 8 oz/240 mL of malt liquor (7% alcohol), 5 oz/150 mL of wine (12% alcohol), or 1.5 oz/45 mL of distilled spirits (40% alcohol);
13. Poor blood pressure control is indicated after treatment by a systolic pressure greater than 160 mmHg or diastolic pressure greater than 100 mmHg during screening;
14. Pregnancy, planned pregnancy, lactation;
15. Treatment with any other investigational therapy or device within 30 days or within 5 half-lives, whichever is longer, prior to screening;
16. Mental instability or incompetence that may compromise the validity of informed consent or ability to adhere to study requirements;
17. Any other condition(s) that would compromise the safety of the patient or compromise the quality of the clinical study, as judged by the investigator.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-12-09 (Estimated); Study Completion 2028-01-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who achieve the composite response criteria at Week 52 | Baseline to week 52 .
  1. ALP < 1.67×ULN
  2. and ALP decrease of ≥15%
  3. and TB ≤1.0× ULN

SECONDARY OUTCOMES:
Response to treatment based on γ-glutamyl transpeptidase (GGT) normalization in patients with baseline GGT>1.0× ULN at Week 26 and Week 52 | Basline to week 26 and week 52 .
Response to treatment based on alanine aminotransferase (ALT) normalization in patients with baseline ALT >1.0× ULN at Week 26 and Week 52 | Basline to week 26 and week 52 .
Proportion of patients with ALP< 1.67× ULN and TB ≤1.0× ULN and ALP decrease of ≥15% from baseline at Week 26 | Baseline to week 26 .
Response to treatment based on AST normalization in patients with baseline AST>1.0× ULN at Week 26 and Week 52 | Baseline to week 26 and week 52 .
Proportion of patients with ALP≤ 3× ULN and AST ≤ 2 × ULN and TB≤ 1.0×ULN at Week 52 | Baseline to week 52 .
The first occurrence of clinical outcome events as defined | up to 56 weeks
  Overall death Liver transplantation Model for End-Stage Liver Disease (MELD)-Na score >14 for at least 2 consecutive visits Ascites requiring treatment
  Hospitalization for new onset or recurrence of any of the following:
  i. Variceal bleeding
  ii. Hepatic encephalopathy (as defined by a West Haven score ≥2)
  iii. Spontaneous bacterial peritonitis (confirmed by culture from diagnostic paracentesis).
Assessment of treatment-emergent AEs (TEAEs) | up to 56 weeks
  Safety

OTHER OUTCOMES:
Absolute changes of liver stiffness measured by iLivTouch | week 26, week 52

CONTACTS AND LOCATIONS:
Overall Officials: Ma Xiong, MD, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (41):
- China (41):
  - The First Affiliated Hospital of USTC Anhui Provincial Hospital, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Mengchao Hepatobiliary Hospital Of Fujian Medical University, Fuzhou, Fujian
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen Third People's Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hebei Medical University Third Hospital, Shijiazhuang, Hebei
  - The Fourth Hospital Of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Taihe Hospital of Shiyan, Shiyan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - The Fifth People's Hospital of Suzhou, Suzhou, Jiangsu
  - The Fifth People's Hospital Of Wuxi, Wuxi, Jiangsu
  - The Third People's Hospital of Zhenjiang, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Sixth People's Hospital of Shenyang, Shenyang, Liaoning
  - Baoji People's Hospital, Baoji, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Linyi People's Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Shanghai Jiao Tong University School of Medicine Ruijin Hospital, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiliated To Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - Hangzhou Xixi Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang